CLINICAL TRIAL: NCT00745069
Title: 4-Week Randomized Multicenter DB, Placebo- and Active-controlled, Parallel-group, Forced-titration Phase 2B Study of Efficacy and Safety With CG5503 Prolonged Release (PR) to 233 mg BID and Oxycodone PR to 20 mg BID vs Placebo in Subjects With Moderate to Severe Chronic Pain of Knee Osteoarthritis
Brief Title: Efficacy and Safety of Tapentadol Extended Release Tablets in the Treatment of Moderate to Severe Pain in Subjects With Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004183
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Osteoarthitis; Chronic Pain; Knee Pain
Keywords: Tapentadol; Osteoarthritis; Analgesia; Chronic pain
MeSH Terms: conditions — Chronic Pain; Osteoarthritis; Agnosia | interventions — Tapentadol

INTERVENTIONS:
Drug: tapentadol HCl

SUMMARY:
The purpose of this study was to examine a low and high dose of tapentadol extended release tablet taken orally twice a day to reduce pain in subjects suffering from chronic moderate to severe pain due to osteoarthritis of the knee during a 4-week period. Subjects steadily increased their dose up to the low (100 mg) or high (200 mg) dose. Pain relief was compared to subjects taking placebo tablets or oxycodone extended release tablet, 20 mg. The serum concentrations and safety of tapentadol and oxycodone were also examined.

DETAILED DESCRIPTION:
Arthritis is the most common chronic debilitating disease in the United States (more than 43 million people or 1 in 6). Osteoarthritis of the knee is a very common and a major cause of disability. Pharmacological treatment includes the following analgesics: non-steroidal anti-inflammatory drugs (NSAIDs), cyclo-oxygenase II (COX-II) inhibitors, acetaminophen and opioids. Despite the numerous available analgesic medications, 60% to 80% of patients suffering from chronic pain are currently treated inadequately. Opioid analgesics have been shown to be efficacious in chronic non-malignant pain and can be an important therapeutic asset. The study was a 4-week randomized multicenter double-blind, placebo- and active-controlled, parallel-group, forced-titration phase 2B study of efficacy and safety with tapentadol extended release (ER) to 233 mg BID and oxycodone PR to 20 mg BID vs placebo in subjects with moderate to severe chronic pain of knee osteoarthritis. Primary efficacy outcome was the average pain intensity 24 hours before the last evaluation time or 29 days. Safety was evaluated by reporting of adverse events, laboratory tests, vital sign measures, ECGs. This study hypothesis was that tapentadol extended release was effective in relieving chronic moderate to severe pain from knee osteoarthritis compared to treatment with placebo using 2 dosing regimens for tapentadol.

tapentadol extended release white, fim-coated tablet taken orally twice a day during a 4-week period at a dose that steadily increased up to 100 mg or 200 mg; placebo tablets; or oxycodone extended release tablet, 20 mg.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a clinical diagnosis of osteoarthritis of the knee based symptoms and/or radiographic criteria present for at least 3 months
* Moderate to severe chronic pain due to knee osteoarithritis

Exclusion Criteria:

* Previously opioid treated subject who had a history of withdrawal after cessation of the opioid
* History of seizure disorder, psychiatric disease and history of head trauma requiring evaluation by hospital based staff, or unconsciousness of unknown origin. Subjects who, in the investigator's judgment, have well-controlled depression or anxiety disorder may participate
* Subjects with history of uncontrolled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 95 mmHg)
* Intake of tricyclic antidepressants, serotonin norepinephrine reuptake inhibitors, barbiturates, neuroleptics, monoamine oxidase inhibitors, and antiparkinsonian drugs within the 30 days prior to the screening visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Actual)
Dates: Start 2004-07; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Average pain intensity over the preceding 24 hours evaluated at the last timepoint or 29 days using a visual scale.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index at the last timepoint or 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Eichenbaum G, Gohler K, Etropolski M, Steigerwald I, Pergolizzi J, Kim M, Vorsanger G. Does tapentadol affect sex hormone concentrations differently from morphine and oxycodone? An initial assessment and possible implications for opioid-induced androgen deficiency. J Opioid Manag. 2015 May-Jun;11(3):211-27. doi: 10.5055/jom.2015.0270. PMID 25985806
- See also: Efficacy and safety of tapentadol extended release tablets in the treatment of moderate to severe pain in subjects with knee osteoarthritis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=561&filename=CR004183_CSR.pdf